CLINICAL TRIAL: NCT06356311
Title: A Phase 3, Multicenter, Open-label, Randomized Study to Compare the Efficacy and Safety of MK-2870 Versus Treatment of Physician's Choice in 3L+ Advanced/Metastatic Gastroesophageal Adenocarcinoma (Gastric Adenocarcinoma, Gastroesophageal Junction Adenocarcinoma, and Esophageal Adenocarcinoma)
Brief Title: A Study to Evaluate Sacituzumab Tirumotecan (MK-2870) in Advanced/Metastatic Gastroesophageal Adenocarcinoma (MK-2870-015)
Acronym: TroFuse-015
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2870-015; 2023-505423-31-00 (Registry Identifier: EU CT); U1111-1291-7109 (Registry Identifier: UTN); MK-2870-015 (Other: MSD Id); jRCT2031240133 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Gastroesophageal Cancer
Keywords: Gastroesophageal cancer; Gastroesophageal adenocarcinoma; Gastric adenocarcinoma; Esophageal adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — trifluridine tipiracil drug combination; Irinotecan; Paclitaxel; Docetaxel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sacituzumab tirumotecan (Experimental): Participants will receive sacituzumab tirumotecan at a dose of 4mg/kg by intravenous (IV) infusion on days 1, 15, and 29 of every 42-day cycle.
  Interventions: Biological: Sacituzumab tirumotecan; Drug: Rescue medication; Drug: Supportive care measures
- Treatment of Physician's Choice (TPC) (Active Comparator): TPC include either trifluridine-tipiracil (35 mg/m^2 orally (PO) twice a day (BID) on days 1 to 5 and 8 to 12 of every 28-day cycle), irinotecan (150 mg/m^2 IV on days 1 and 15 of every 28-day cycle), paclitaxel (80 mg/m^2 IV on days 1, 8, and 15 of every 28-day cycle), or docetaxel (75 mg/m^2 IV on day 1 of every 21-day cycle).
  Interventions: Drug: Trifluridine-Tipiracil; Drug: Irinotecan; Drug: Paclitaxel; Drug: Docetaxel; Drug: Supportive care measures

INTERVENTIONS:
Biological: Sacituzumab tirumotecan — Participants will receive sacituzumab tirumotecan as 4mg/kg IV infusion on days 1, 15, and 29 of every 42-day cycle.
  Other Names: SKB264. MK-2870
  Arms: Sacituzumab tirumotecan
Drug: Trifluridine-Tipiracil — Trifluridine-tipiracil will be administered at 35 mg/m^2 as tablet orally twice a day on days 1-5 and 8-12 of every 28-day cycle.
  Arms: Treatment of Physician's Choice (TPC)
Drug: Irinotecan — Irinotecan will be administered at a dose of 150 mg/m^2 by IV infusion on days 1 and 15 of every 28-day cycle.
  Arms: Treatment of Physician's Choice (TPC)
Drug: Paclitaxel — Paclitaxel will be administered at a dose of 80 mg/m^2 by IV infusion on days 1, 8 and 15 of every 28-day cycle.
  Arms: Treatment of Physician's Choice (TPC)
Drug: Docetaxel — Docetaxel will be administered at a dose of 75 mg/m^2 by IV infusion on day 1 of a 21-day cycle.
  Arms: Treatment of Physician's Choice (TPC)
Drug: Rescue medication — Participants are allowed to take rescue medication for stomatitis or oral mucositis. At the discretion of the investigator, participants are provided with a prescription for rescue medications. Recommended rescue medications are antihistamine, histamine-2 (H2) receptor antagonist, acetaminophen or equivalent, dexamethasone or equivalent infusion or steroid mouthwash (dexamethasone or equivalent), antiemetic medications, oral nystatin suspension or antifungal medications, antidiarrheal agents, antiemetic agents, opiate and non-opiate analgesic agents, appetite stimulants, and granulocyte and erythroid growth factors.
  Arms: Sacituzumab tirumotecan
Drug: Supportive care measures — Participants are allowed to take supportive care measures for the management of adverse events associated with study intervention at the discretion of the investigator. Supportive care measures may include but are not limited to antidiarrheal agents, antiemetic agents, opiate and non-opiate analgesic agents, appetite stimulants, and granulocyte and erythroid growth factors.

SUMMARY:
This study will compare how safe and effective sacituzumab tirumotecan is versus the treatment of physician's choice (TPC) in participants with advanced/metastatic gastroesophageal adenocarcinoma. The primary hypothesis of this study is sacituzumab tirumotecan is superior to TPC with respect to Overall Survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically-or cytologically-confirmed diagnosis of advanced, unresectable or metastatic gastric adenocarcinoma, gastroesophageal junction adenocarcinoma, or esophageal adenocarcinoma
* Has measurable disease per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) as assessed by the local site investigator/radiology. Lesions situated in a previously-irradiated area are considered measurable if progression has been shown in such lesions.
* Has received, and progressed on, at least 2 prior chemotherapy and/or immunotherapy regimens for advanced, unresectable or metastatic gastroesophageal adenocarcinoma.
* Participants are eligible regardless of human epidermal growth factor receptor-2 (HER2) status. Participants who are HER2+ must have previously received trastuzumab where available/appropriate
* Has adequate organ function
* Has provided tumor tissue sample for determination of trophoblast cell-surface antigen 2 (TROP2) status by the central laboratory before randomization for stratification
* Participants who have AEs due to previous anticancer therapies must have recovered to Grade ≤1 or baseline (except for alopecia and vitiligo). Participants with endocrine related AEs who are adequately treated with hormone replacement therapy are eligible
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 3 days before randomization
* Has ability to swallow oral medication for those who may receive trifluridine-tipiracil
* Human immunodeficiency virus (HIV)-infected participants must have well-controlled HIV on antiretroviral therapy (ART)
* Hepatitis B surface antigen (HBsAg)-positive participants are eligible if they have received hepatitis B virus (HBV) antiviral therapy and have undetectable HBV viral load
* Participants with a history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable

Exclusion Criteria:

* Has a history of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or severe corneal disease that prevents/delays corneal healing
* Has Grade ≥2 peripheral neuropathy
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous history of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis, or chronic diarrhea)
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, uncontrolled symptomatic arrhythmia, prolongation of corrected QT interval (QTcF) to >480 ms, and/or other serious cardiovascular and cerebrovascular diseases within 6 months before the first dose of study intervention
* Has accumulation of pleural, ascitic, or pericardial fluid requiring drainage or diuretic drugs within 2 weeks before the first dose of study intervention
* Has received prior treatment with a trophoblast antigen 2(TROP2) targeted antibody-drug conjugate (ADC), a topoisomerase 1 inhibitor based, and/or a topoisomerase 1 inhibitor-based chemotherapy.
* Has received prior systemic anticancer therapy within 2 weeks before the first dose of study intervention
* Has received prior radiotherapy within 2 weeks before the first dose of study intervention, has radiation-related toxicities, requiring corticosteroids, and/or has had radiation pneumonitis
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Is currently receiving a strong and/or moderate inducer/inhibitor of cytochrome P450 3A4 (CYP3A4) that cannot be discontinued for the duration of treatment with study intervention. The required washout period before starting study intervention is 2 weeks
* Has received an investigational agent or has used an investigational device within 4 weeks before the first dose of study intervention
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has an active infection requiring systemic therapy
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castlemans's Disease
* Has concurrent active hepatitis B (defined as hepatitis B surface antigen (HBsAg) positive and/or detectable HBV deoxyribonucleic acid (DNA)) and Hepatitis C virus (HCV) defined as anti-HCV antibody (Ab) positive and detectable HCV ribonucleic acid (RNA)) infection
* Has had major surgery or significant traumatic injury within 4 weeks before the first dose of study intervention. Anticipation of the need for major surgery during the course of treatment with study intervention is also exclusionary
* Has severe hypersensitivity (Grades >=3) to the study interventions, any of their excipients, and/or to another biologic therapy
* Has a history of (noninfectious) pneumonitis/ interstitial lung disease (ILD) that required steroids or has current pneumonitis/ILD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2027-01-04 (Estimated); Study Completion 2027-05-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to ~ 31 months
  OS is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to ~ 25 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1). PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by blinded independent central review (BICR) will be presented.
Objective Response Rate (ORR) | Up to ~ 25 months
  ORR is defined as the percentage of participants with CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience CR or PR as assessed by BICR will be presented.
Duration of Response (DOR) | Up to ~ 25 months
  For participants who demonstrate a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until PD or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Number of Participants Who Experience an Adverse Event (AE) | Up to ~ 36 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Number of Participants Who Discontinue Study Intervention Due to an AE | Up to ~ 36 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (168):
- United States (17):
  - Banner MD Anderson Cancer Center ( Site 0119), Gilbert, Arizona
  - UCLA Hematology/Oncology - Santa Monica ( Site 0140), Los Angeles, California
  - AdventHealth Orlando-AdventHealth Medical Group Hematology & Oncology at Orlandoc ( Site 0129), Orlando, Florida
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital-Research ( Site 0108), Marietta, Georgia
  - University of Chicago Medical Center ( Site 0120), Chicago, Illinois
  - University of Kentucky Chandler Medical Center-Medical Oncology ( Site 0124), Lexington, Kentucky
  - The University of Louisville, James Graham Brown Cancer Center-James Graham Brown Cancer Center ( Site 0113), Louisville, Kentucky
  - Norton Audubon Hospital-Norton Cancer Institute - Audubon ( Site 0105), Louisville, Kentucky
  - Henry Ford Hospital ( Site 0107), Detroit, Michigan
  - Sanford Fargo Medical Center-Roger Maris Cancer Center ( Site 0138), Fargo, North Dakota
  - Oregon Health and Science University ( Site 0104), Portland, Oregon
  - UPMC Hillman Cancer Center ( Site 0126), Pittsburgh, Pennsylvania
  - MUSC Hollings Cancer Center-Hematology Oncology ( Site 0122), Charleston, South Carolina
  - Sanford Cancer Center ( Site 0136), Sioux Falls, South Dakota
  - The West Clinic, PLLC dba West Cancer Center ( Site 0110), Germantown, Tennessee
  - Inova Schar Cancer ( Site 0106), Fairfax, Virginia
  - Fred Hutchinson Cancer Center ( Site 0111), Seattle, Washington
- Belgium (4):
  - Institut Jules Bordet-GastroIntestinal Medical Oncology ( Site 1003), Anderlecht, Bruxelles-Capitale, Region de
  - Cliniques universitaires Saint-Luc-Medical Oncology ( Site 1001), Brussels, Bruxelles-Capitale, Region de
  - UZ Leuven-Digestive Oncology ( Site 1000), Leuven, Vlaams-Brabant
  - AZ Delta vzw ( Site 1002), Roeselare, West-Vlaanderen
- Brazil (9):
  - Centro de Pesquisa Clínica do Instituto do Câncer do Ceará ( Site 0405), Fortaleza, Ceará
  - Liga Norte Riograndense Contra o Câncer-Centro de Pesquisa Clínica ( Site 0406), Natal, Rio Grande do Norte
  - Hospital de Caridade de Ijuí ( Site 0412), Ijuí, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceição-Centro Integrado de Pesquisa em Oncologia ( Site 0400), Porto Alegre, Rio Grande do Sul
  - Centro de Hematologia e Oncologia ( Site 0404), Joinville, Santa Catarina
  - Fundação Pio XII - Hospital de Câncer de Barretos-Unidade de Pesquisa Clínica ( Site 0401), Barretos, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto ( Site 0411), São José do Rio Preto, São Paulo
  - A. C. Camargo Cancer Center ( Site 0409), São Paulo
  - IBCC - Núcleo de Pesquisa e Ensino ( Site 0402), São Paulo
- McGill University Health Centre ( Site 0201), Montreal, Quebec, Canada
- Chile (5):
  - Centro de Estudios Clínicos SAGA-CECSAGA ( Site 0503), Santiago, Region M. de Santiago
  - FALP-UIDO ( Site 0500), Santiago, Region M. de Santiago
  - Clínica UC San Carlos de Apoquindo-Hemato-Oncology ( Site 0502), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 0501), Santiago, Region M. de Santiago
  - James Lind Centro de Investigacion del Cancer ( Site 0506), Temuco, Región de la Araucanía
- China (33):
  - Anhui Provincial Cancer Hospital-medical oncology ( Site 3016), Hefei, Anhui
  - Second Affiliated hospital of Anhui Medical University-Oncology ( Site 3038), Hefei, Anhui
  - Chongqing University Three Gorges Hospital ( Site 3036), Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital ( Site 3007), Fuzhou, Fujian
  - The 900th Hospital of the Joint Logistics Support Force of PLA ( Site 3008), Fuzhou, Fujian
  - The First Affiliated hospital of Xiamen University-oncology ( Site 3011), Xiamen, Fujian
  - Zhongshan Hospital Affiliated to Xiamen University ( Site 3013), Xiamen, Fujian
  - Sun Yat-Sen University Cancer Center ( Site 3001), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital-Department of Oncology ( Site 3019), Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College ( Site 3034), Shantou, Guangdong
  - Affiliated Cancer Hospital of Guangxi Medical University ( Site 3047), Nanning, Guangxi
  - Fourth Hospital of Hebei Medical University ( Site 3015), Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital-Harbin Medical University Cancer Hospital ( Site 3005), Harbin, Heilongjiang
  - Henan Cancer Hospital-henan cancer hospital ( Site 3002), Zhengzhou, Henan
  - Hubei Cancer Hospital ( Site 3012), Wuhan, Hubei
  - Xiangyang Central Hospital ( Site 3045), Xiangyang, Hubei
  - Hunan Cancer Hospital ( Site 3014), Changsha, Hunan
  - The First Affiliated Hospital of Soochow University ( Site 3040), Suzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University-Oncology Department ( Site 3037), Nanchang, Jiangxi
  - Jilin Province Tumor Hospital ( Site 3018), Changchun, Jilin
  - LinYi Cancer Hospital-Gastrology department ( Site 3024), Linyi, Shandong
  - Fudan University Shanghai Cancer Center-medical oncology ( Site 3009), Shanghai, Shanghai Municipality
  - Zhongshan Hospital,Fudan University-Oncology ( Site 3003), Shanghai, Shanghai Municipality
  - Renji Hosp,Shanghai Jiao Tong University School of Medicine ( Site 3042), Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University ( Site 3035), Chengdu, Sichuan
  - Sichuan Cancer hospital. ( Site 3030), Chengdu, Sichuan
  - Beijing Anzhen Nanchong Hospital of Capital Medical University (Nanchong Central Hospital) ( Site 3029), Nanchong, Sichuan
  - Xinjiang Medical University Cancer Hospital - Urumchi-The No.11 of Surgery building ( Site 3010), Ürümqi, Xinjiang
  - Yunnan Province Cancer Hospital ( Site 3031), Kunming, Yunnan
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine-Oncology ( Site 3006), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital-Oncology ( Site 3021), Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province ( Site 3020), Linhai, Zhejiang
  - Yueqing People's Hospital ( Site 3041), Yueqing, Zhejiang
- Colombia (5):
  - Centro Cancerológico del Caribe (CECAC) ( Site 0606), Barranquilla, Atlántico
  - FUNDACION CTIC CENTRO DE TRATAMIENTO E INVESTIGACION SOBRE CANCER LUIS CARLOS SARMIENTO ANGULO ( Site 0602), Bogotá, Bogota D.C.
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia-Center Investigator ( Site 0603), Bogotá, Bogota D.C.
  - Sociedad de Oncología Y Hematología del Cesar S.A.S. ( Site 0600), Valledupar, Cesar Department
  - Fundación Valle del Lili-Fundacion Valle del Lili ( Site 0607), Cali, Valle del Cauca Department
- Denmark (3):
  - Rigshospitalet ( Site 1102), Copenhagen, Capital Region
  - Aalborg Universitetshospital, Syd-Department of Oncology ( Site 1103), Aalborg, North Denmark
  - Odense Universitetshospital-Department of oncology ( Site 1101), Odense, Region Syddanmark
- France (9):
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cance-Medical Oncology ( Site 1211), Bordeaux, Aquitaine
  - CENTRE LEON BERARD-Medical oncology ( Site 1208), Lyon, Auvergne-Rhône-Alpes
  - Centre François Baclesse ( Site 1202), Caen, Calvados
  - CHU Rangueil-Digestive oncology department ( Site 1210), Toulouse, Haute-Garonne
  - Centre Oscar Lambret ( Site 1206), Lille, Hauts-de-France
  - Centre Eugène Marquis Rennes - Centre de Lutte Contre le Cancer ( Site 1203), Rennes, Ille-et-Vilaine
  - Centre Hospitalier Universitaire de Poitiers ( Site 1209), Poitiers, Vienne
  - Hôpital Saint-Louis ( Site 1201), Paris
  - Institut Mutualiste Montsouris-Oncology ( Site 1216), Paris, Île-de-France Region
- Germany (6):
  - NCT-Department of Medical Oncology ( Site 1302), Heidelberg, Baden-Wurttemberg
  - Universitätsmedizin Göttingen - Georg-August-Universität ( Site 1310), Göttingen, Lower Saxony
  - Universitaetsklinikum Carl Gustav Carus Dresden-Medical Dept I - Medical Oncology ( Site 1307), Dresden, Saxony
  - Städtisches Krankenhaus Kiel-2. Medizinische Klinik ( Site 1306), Kiel, Schleswig-Holstein
  - Charité Campus Virchow-Klinikum-Klinik Hämatologie Onkologie Tumorimmunologie ( Site 1304), Berlin
  - Facharztzentrum Eppendorf-Facharztzentrum Eppendorf ( Site 1300), Hamburg
- Hong Kong (3):
  - Queen Mary Hospital ( Site 3100), Hong Kong
  - Prince of Wales Hospital ( Site 3102), Shatin
  - Queen Elizabeth Hospital ( Site 3101), Yau Ma Tei
- Israel (5):
  - Hillel Yaffe Medical Center ( Site 1604), Hadera
  - Rambam Health Care Campus-Oncology Division ( Site 1600), Haifa
  - Hadassah Medical Center ( Site 1603), Jerusalem
  - Rabin Medical Center ( Site 1605), Petah Tikva
  - Sourasky Medical Center ( Site 1602), Tel Aviv
- Italy (5):
  - Azienda Ospedaliera Universitaria dell'Università "Luigi Van-UOC Oncoematologia ( Site 1704), Napoli, Campania
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS -Medical Oncology ( Site 1703), Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 1700), Milan, Lombardy
  - Azienda Ospedaliero Universitaria Pisana ( Site 1702), Pisa, Tuscany
  - Ospedale San Raffaele-Oncologia Medica ( Site 1701), Milan
- Japan (8):
  - Aichi Cancer Center ( Site 3307), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 3300), Kashiwa, Chiba
  - Kochi Medical School Hospital ( Site 3304), Nankoku, Kochi
  - Saitama Prefectural Cancer Center ( Site 3302), Kitaadachi-gun, Saitama
  - National Cancer Center Hospital ( Site 3301), Chūō, Tokyo
  - Cancer Institute Hospital of JFCR ( Site 3306), Koto, Tokyo
  - National Hospital Organization Kyushu Cancer Center ( Site 3303), Fukuoka
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute ( Site 3305), Osaka
- Malaysia (5):
  - Hospital Pulau Pinang ( Site 3403), George Town, Pulau Pinang
  - National Cancer Institute-Radiotherapy and Oncology ( Site 3404), Putrajaya, Putrajaya
  - Sarawak General Hospital-Radiotherapy Unit ( Site 3401), Kuching, Sarawak
  - University Malaya Medical Centre-Clinical Oncology ( Site 3402), Kuala Lumpur
  - Pantai Hospital Kuala Lumpur-Cancer Centre ( Site 3408), Kuala Lumpur
- Mexico (6):
  - CANCER TREAMTENT CLINIC AND CLINICAL TRIALS SA DE CV ( Site 0814), Guadalajara, Jalisco
  - COI Centro Oncologico Internacional S.A.P.I. de C.V.-Investigation Unit COI ( Site 0802), Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran-Oncologia y Hematologia ( Site 0805), Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez"-Servicio de Oncología ( Site 0809), Monterrey, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca ( Site 0810), Oaxaca City, Oaxaca
  - Centro Potosino de Investigación Médica ( Site 0801), San Luis Potosí City, San Luis Potosí
- Peru (6):
  - Instituto Regional de Enfermedades Neoplasicas del Centro (IREN CENTRO) ( Site 0904), Concepción, Departamento de Junín
  - Hospital de Alta Complejidad La Libertad-Unidad de Investigación en Oncología ( Site 0902), Trujillo, La Libertad
  - Clínicas AUNA Sede Chiclayo ( Site 0907), Chiclayo, Lambayeque
  - Clínica Internacional - Sede San Borja ( Site 0906), Lima
  - IPOR Instituto Peruano de Oncología & Radioterapia-Centro de Investigación ( Site 0905), Lima
  - INSTITUTO NACIONAL DE ENFERMEDADES NEOPLASICAS-Medical Oncology ( Site 0900), Lima
- Poland (6):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 1807), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Onkologii i Radioterapii ( Site 1800), Warsaw, Masovian Voivodeship
  - Bialostockie Centrum Onkologii ( Site 1804), Bialystok, Podlaskie Voivodeship
  - Szpitale Pomorskie Sp. z o. o.-Oddział Onkologii Klinicznej " Profil Jednego Dnia " ( Site 1810), Gdynia, Pomeranian Voivodeship
  - Szpital Wojewódzki w Koszalinie. ( Site 1801), Poland, West Pomeranian Voivodeship
  - Swietokrzyskie Centrum Onkologii, Samodzielny Publiczny Zaklad Opieki Zdrowotnej ( Site 1811), Kielce, Świętokrzyskie Voivodeship
- South Korea (6):
  - Seoul National University Bundang Hospital ( Site 3504), Seongnam, Kyonggi-do
  - Seoul National University Hospital-Oncology ( Site 3503), Seoul
  - Severance Hospital, Yonsei University Health System-Medical oncology ( Site 3500), Seoul
  - Asan Medical Center-Department of Oncology ( Site 3501), Seoul
  - Samsung Medical Center-Division of Hematology/Oncology ( Site 3502), Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital ( Site 3505), Seoul
- Spain (6):
  - Hospital Universitario Marqués de Valdecilla ( Site 1901), Santander, Cantabria
  - CHUAC-Complejo Hospitalario Universitario A Coruña ( Site 1905), A Coruña, La Coruna
  - COMPLEJO HOSPITALARIO DE NAVARRA-Medical Oncology ( Site 1904), Pamplona, Navarre
  - Hospital Universitario Central de Asturias-Medical Oncology ( Site 1902), Oviedo, Principality of Asturias
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 1900), Barcelona
  - Hospital Clinico San Carlos ( Site 1903), Madrid
- Taiwan (5):
  - China Medical University Hospital ( Site 3603), Taichung
  - National Cheng Kung University Hospital-Clinical Trial Center ( Site 3604), Tainan
  - National Taiwan University Hospital ( Site 3600), Taipei
  - Taipei Veterans General Hospital ( Site 3601), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 3602), Taoyuan District
- Thailand (3):
  - Chulalongkorn University ( Site 3702), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital ( Site 3700), Bangkok, Bangkok
  - Songklanagarind hospital ( Site 3701), Hat Yai, Changwat Songkhla
- Turkey (Türkiye) (8):
  - Baskent University Dr. Turgut Noyan Research and Training Center-ONCOLOGY ( Site 2104), Adana
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 2100), Ankara
  - Ankara Bilkent Şehir Hastanesi-Medical Oncology ( Site 2101), Ankara
  - Dicle Üniversitesi-oncology ( Site 2108), Diyarbakır
  - Atatürk Üniversitesi-onkoloji ( Site 2111), Erzurum
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 2106), Istanbul
  - Samsun Medical Park Hastanesi-medical oncology ( Site 2110), Samsun
  - Yuzuncu Yil University Dursun Odaba Tp Merkezi-Medical Oncology ( Site 2109), Van
- United Kingdom (4):
  - Addenbrooke's Hospital ( Site 2203), Cambridge, Cambridgeshire
  - Ninewells Hospital and Medical School-Oncology Petty ( Site 2209), Dundee, Dundee City
  - St Bartholomew's Hospital ( Site 2206), London, London, City of
  - The Christie NHS Foundation Trust-Medical Oncology ( Site 2201), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26288&tenant=MT_MSD_9011